CLINICAL TRIAL: NCT07280325
Title: Moxie: A Self-management Education and Support Program Using Advertising Principles to Reduce Rehospitalization for Cardiovascular-related Illnesses
Brief Title: Moxie Self-Management and Education Support Program
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Emergence Creative (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: Pro00141473
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-09

CONDITIONS: Chronic Kidney Disease; Diabetes (DM); Heart Disease; Stroke; Chronic Disease
Keywords: Chronic Disease Self-Management; Pragmatic Trial; Chronic Disease Education
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus; Heart Diseases; Stroke; Chronic Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Moxie SMES Program (Experimental): Participants randomized to this arm receive weekly mailers for the Moxie SMES Program and an invitation to participate in the digital health component.
  Interventions: Behavioral: Moxie SMES Letters
- Facilitated Relay (Experimental): Participants randomized to this arm receive a one-time facilitated relay letter to share with their pharmacist and primary care provider.
  Interventions: Behavioral: Facilitated Relay Letter
- Moxie SMES Program and Facilitated Relay (Experimental): Participants randomized to this arm receive weekly mailers for the Moxie SMES Program, an invitation to participate in the digital health component, and the one-time facilitated relay letter to share with their pharmacist and primary care provider.
  Interventions: Behavioral: Moxie SMES Letters; Behavioral: Facilitated Relay Letter
- Control (No Intervention): Participants randomized to this arm receive standard of care only.

INTERVENTIONS:
Behavioral: Moxie SMES Letters — Weekly mailer for the Moxie SMES Program.
  Arms: Moxie SMES Program; Moxie SMES Program and Facilitated Relay
Behavioral: Facilitated Relay Letter — One-time Facilitated Relay letter for the participant to share with their healthcare provider.
  Arms: Facilitated Relay; Moxie SMES Program and Facilitated Relay

SUMMARY:
Health education and self-management support are key facilitators of health behaviours. Moxie is a mixed media, self-management, education and support program for Albertans living with cardiovascular-related chronic conditions. Moxie is built upon our previous work within the ACCESS study (2015-21, n=4761), a RCT that previously tested the Moxie intervention in Alberta. Results demonstrated that MOXIE reduced the rate of hospitalizations (notably for hypertension, angina, hyper/hypoglycemia, heart failure decompensation, and acute kidney complications) by 34% in a population of low-income seniors living with cardiovascular-related chronic conditions.

However, before Moxie can be effectively implemented province-wide, another trial is necessary to determine whether benefits can be observed in a larger cohort of patients with cardiovascular-related chronic conditions recruited immediately after hospital discharge (n=9000). Furthermore, the effectiveness of the two components of the ACCESS trial intervention will be assessed individually:

(a) The Moxie Program, a tailored health and disease education component developed by a user-experience-centric design process incorporating patients, behavioural scientists, disease specialists, health system administrators and marketing/advertising professionals; and (b) the facilitated relay of clinical information to healthcare providers (letters).

The trial is designed as a 2x2 factorial pragmatic, individual-level randomized pragmatic trial of these different interventions. This would yield the following groups:

1. Moxie SMES Program
2. Facilitated Relay
3. Moxie SMES Program and Facilitated Relay
4. True control

Self-management education and support (SMES) intervention: This includes weekly physical mailers sent directly to patients' homes throughout the study containing information about chronic conditions, medication use, diet, physical activity, smoking cessation, and self-management/wellness principles. These messages will be refined by the social impact creative design partner and reviewed by clinicians and patients to ensure clinical safety and appropriate tone. Weekly mailers will encourage participants to enroll and consent to participate in the digital program by scanning a QR code or accessing a website where they will sign up for their own personalized Moxie mobile health app, complete a digital consent form and opt-in for electronic delivery of Moxie messages.

Facilitated relay intervention: Participants allocated to this intervention will receive letters by mail, one addressed to them, one to their primary care provider, and one to their pharmacist. The letters will not be sent to their primary care provider directly; rather, they will be sent to patients who will be encouraged to take them to their primary care provider and pharmacist should they decide to do so. We hope this will empower patients to start discussions with their healthcare providers. This also supports patient autonomy by enabling patients to decide whether they want to take them to their provider or not. If for whatever reason they do not feel that this is going to be beneficial or of interest, they are not required to do so. The letter would contain a note to the patient's healthcare provider stating that their patient is at-risk of cardiovascular disease and that evidence has shown that the pharmacotherapy is effective in improving outcomes for patients similar to the participant.

The primary outcome is readmission for cardiovascular-specific ambulatory care-sensitive conditions (ACSC) based on the most responsible diagnosis listed in CIHI Discharge Abstract Database-(DAD), using established algorithms within 12 months from randomization. This outcome includes all repeat admissions in the study period as recorded in the health record. This outcome is a count variable. We will calculate and compare each intervention arm's mean number and distribution of hospitalizations.

ELIGIBILITY:
Inclusion Criteria:

Eligible participants will be adults aged 40-85 years who are being discharged to their home from general internal medicine or family medicine inpatient services (hospitalist) in one of 10 Alberta acute care facilities, whose admitting diagnosis was diabetes, coronary artery disease, heart failure, chronic kidney disease, or hypertension (see appendix for list of inclusion diagnoses).

Exclusion Criteria:

Individuals who live at the same address/household as a person who is already in the study and/or those discharged from hospitals to continuing care facilities, rehabilitation facilities or another hospital will not be eligible to take part in the study. Individuals whose goals of care at the time of discharge from acute care were oriented towards comfort (i.e. C1 or C2 Goals of Care) will not be eligible to take part in the study. Individuals with markers indicating lack of competency/capacity in their inpatient ConnectCare record such as anything but full capacity on the medical record (i.e. "incapacitated" or "needs review"), or presence of an alternative decision maker, agent, or legal guardian listed on the medical record.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9000 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Hospital Readmissions | Within 12 months from randomization.
  Readmission for cardiovascular-specific ambulatory care-sensitive conditions (ACSC) based on the most responsible diagnosis listed in CIHI-DAD (23). This outcome includes all repeat admissions in the study period as recorded in the AHS record that is sent to CIHI for inclusion in the Discharge Abstract Database (DAD). This outcome is a count variable. We will calculate and compare each intervention arm's mean number and distribution of hospitalizations.

SECONDARY OUTCOMES:
Overall Mortality | Within 12 months of randomization.
  Death, for the purpose of this study, refers to all-cause mortality. The data source for this outcome is the Canadian Vital Statistics Database (CVSD).
Cardiovascular-Kidney-Metabolic Death | Within 12 months from randomization.
  The CVSD also records an ICD-10 code for the most responsible cause of death provided by the most responsible healthcare provider (death in an inpatient facility) or the coroner's office (death in the community). This code can be used to identify those who die of relevant causes if the assigned ICD-10 code is within the following ranges: cardiovascular (I00-I99), diabetes (E10-E14), or kidney-related (N00-N29).
Cardioprotective Medication Initiation | Within 12 months from randomization.
  Using data from Alberta's pharmacy dispensation repository, we will identify when a patient with an indicated condition starts a new medication that they were not previously taking in the prior 12 months. The combination of conditions and medications we will assess for include:
  Heart Failure= ACE/ARB/ARNI, SGLT2 inhibitors, MRA, Statins Chronic kidney disease with proteinuria (no diabetes)= ACE/ARB/ARNI, SGLT2 inhibitors, Statins Chronic kidney disease with proteinuria and diabetes= ACE/ARB/ARNI, SGLT2 inhibitors, Statins, Finerenone Chronic kidney disease without proteinuria= ACE/ARB/ARNI, Statins Coranary artery disease= ACE/ARB/ARNI, Statins Type 2 Diabetes= ACE/ARB/ARNI, SGLT2i or GLP1RA inhibitors, Statins
Medication Adherence | Within 12 months from randomization.
  Adherence to medications such as \ACEi, ARBs, Statins, and other cardioprotective medications listed above will be assessed by calculating the proportion of days covered (calculated using the formula below) (sum of days covered in the period of interest (POI)) ÷ (number of days in the POI) × 100% (24). PDC of 80% or greater is considered adequate adherence. This data is sourced from the Pharmaceutical Information Network, which records information (date, drug name, DIN, strength, quantity, duration) for all dispensed prescriptions from outpatient pharmacies in Alberta.
Primary Care and Specialty Utilization | Within 12 months from randomization.
  Primary care and specialist visits are captured in the Physician Claims Database. Each encounter will be counted as one visit. This outcome is analysed as a count variable. We will calculate and compare the mean number and distribution of primary and specialist care visits.
Healthcare System Costs | Within 12 months from randomization.
  We will include costs for hospitalization and ED visits, physician claims (specialist and primary care physician visit and procedure billing costs), prescription medications, nonphysician ambulatory costs (day medicine and day surgery clinics), and outpatient diagnostic imaging and laboratory costs. The total costs will be calculated as the sum of these costs. Alberta Health uses Canadian Institute of Health Information case-mix grouper methods to estimate hospital costs and ambulatory-case costing methods to estimate emergency department costs. Physician claims will be based on the amount paid by Alberta Health. The cost of medications will be estimated by combining a database containing a comprehensive list of medications dispensed to all Alberta residents with a price list from Alberta Blue Cross, including dispensing fee. Diagnostic imaging and laboratory costs will be based on estimates provided by Alberta Health.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Campbell DJ, Tonelli M, Hemmelgarn B, Mitchell C, Tsuyuki R, Ivers N, Campbell T, Pannu R, Verkerke E, Klarenbach S, King-Shier K, Faris P, Exner D, Chaubey V, Manns B; Interdisciplinary Chronic Disease Collaboration. Assessing outcomes of enhanced chronic disease care through patient education and a value-based formulary study (ACCESS)-study protocol for a 2x2 factorial randomized trial. Implement Sci. 2016 Sep 26;11(1):131. doi: 10.1186/s13012-016-0491-6. PMID 27671037
- [Background] "Statistics Canada Releases New Health of Canadians Report to Summarize the Current State of Health in the Country." Statistics Canadaa, 13 Sept. 2023, www.statcan.gc.ca/en/about/smr09/smr09_142. Accessed 13 Sept. 2023.
- [Background] "A Canadian Peer-reviewed Journal of Population Health and Health Services Research." Statistics Canada, www150.statcan.gc.ca/n1/pub/82-003-x/82-003-x2020010-eng.htm. Accessed 21 Oct. 2020.
- [Background] Sumithira, G., et al. "Incidence and prevalence of diabetes in patients with myocardial infarction: A study in a secondary care hospital." International Journal of Pharmaceutical Research (09752366) 12.3 (2020).
- [Background] Canadian Institute for Health Information. Hospital Morbidity Database (HMDB) metadata. Accessed October 28, 2024.
- [Background] Discharge abstract database metadata. Canadian Institute for Health Information. https://www.cihi.ca/en/dischargeabstract-database-dad-metadata. Published Unknown. Accessed October 17, 2023.
- [Background] "TCPS 2 (2018) - Chapter 3: The Consent Process." Panel on Research Ethics, ethics.gc.ca/eng/tcps2-eptc2_2018_chapter3-chapitre3.html#7b. Accessed 22 Jan. 2020.
- [Background] Ye C, Giangregorio L, Holbrook A, Pullenayegum E, Goldsmith CH, Thabane L. Data withdrawal in randomized controlled trials: Defining the problem and proposing solutions: a commentary. Contemp Clin Trials. 2011 May;32(3):318-22. doi: 10.1016/j.cct.2011.01.016. Epub 2011 Feb 4. PMID 21300179
- [Background] Tripepi G, Jager KJ, Dekker FW, Zoccali C. Selection bias and information bias in clinical research. Nephron Clin Pract. 2010;115(2):c94-9. doi: 10.1159/000312871. Epub 2010 Apr 21. PMID 20407272
- [Background] McCambridge J, Witton J, Elbourne DR. Systematic review of the Hawthorne effect: new concepts are needed to study research participation effects. J Clin Epidemiol. 2014 Mar;67(3):267-77. doi: 10.1016/j.jclinepi.2013.08.015. Epub 2013 Nov 22. PMID 24275499
- [Background] Damschroder LJ, Reardon CM, Widerquist MAO, Lowery J. The updated Consolidated Framework for Implementation Research based on user feedback. Implement Sci. 2022 Oct 29;17(1):75. doi: 10.1186/s13012-022-01245-0. PMID 36309746
- [Background] Eisman AB, Kilbourne AM, Dopp AR, Saldana L, Eisenberg D. Economic evaluation in implementation science: Making the business case for implementation strategies. Psychiatry Res. 2020 Jan;283:112433. doi: 10.1016/j.psychres.2019.06.008. Epub 2019 Jun 7. PMID 31202612
- [Background] Chen W, Qian L, Shi J, Franklin M. Comparing performance between log-binomial and robust Poisson regression models for estimating risk ratios under model misspecification. BMC Med Res Methodol. 2018 Jun 22;18(1):63. doi: 10.1186/s12874-018-0519-5. PMID 29929477
- [Background] Prieto-Merino D, Mulick A, Armstrong C, Hoult H, Fawcett S, Eliasson L, Clifford S. Estimating proportion of days covered (PDC) using real-world online medicine suppliers' datasets. J Pharm Policy Pract. 2021 Dec 29;14(1):113. doi: 10.1186/s40545-021-00385-w. PMID 34965882
- [Background] Jones CL, Jensen JD, Scherr CL, Brown NR, Christy K, Weaver J. The Health Belief Model as an explanatory framework in communication research: exploring parallel, serial, and moderated mediation. Health Commun. 2015;30(6):566-76. doi: 10.1080/10410236.2013.873363. Epub 2014 Jul 10. PMID 25010519
- [Background] Campbell DJT, Tonelli M, Hemmelgarn BR, Faris P, Zhang J, Au F, Tsuyuki RT, Mitchell C, Pannu R, Campbell T, Ivers N, Fletcher J, Exner DV, Manns BJ; Interdisciplinary Chronic Disease Collaboration. Self-Management Support Using Advertising Principles for Older Adults With Low Income at High Cardiovascular Risk: A Randomized Controlled Trial. Circulation. 2023 May 16;147(20):1492-1504. doi: 10.1161/CIRCULATIONAHA.123.064189. Epub 2023 Mar 5. PMID 36871212
- [Background] Shojania KG, McDonald KM, Wachter RM, Owens DK, editors. Closing the Quality Gap: A Critical Analysis of Quality Improvement Strategies (Vol. 1: Series Overview and Methodology). Rockville (MD): Agency for Healthcare Research and Quality (US); 2004 Aug. Report No.: 04-0051-1. Available from http://www.ncbi.nlm.nih.gov/books/NBK43908/ PMID 20734525
- [Background] Campbell DJT, Lee-Krueger RCW, McBrien K, Anderson T, Quan H, Leung AA, Chen G, Lu M, Naugler C, Butalia S. Strategies for enhancing the initiation of cholesterol lowering medication among patients at high cardiovascular disease risk: a qualitative descriptive exploration of patient and general practitioners' perspectives on a facilitated relay intervention in Alberta, Canada. BMJ Open. 2020 Nov 24;10(11):e038469. doi: 10.1136/bmjopen-2020-038469. PMID 33234627
- [Background] McAlister FA, Laupacis A, Armstrong PW. Finding the right balance between precision medicine and personalized care. CMAJ. 2017 Aug 21;189(33):E1065-E1068. doi: 10.1503/cmaj.170107. No abstract available. PMID 28827437
- [Background] Priesterroth L, Grammes J, Holtz K, Reinwarth A, Kubiak T. Gamification and Behavior Change Techniques in Diabetes Self-Management Apps. J Diabetes Sci Technol. 2019 Sep;13(5):954-958. doi: 10.1177/1932296818822998. Epub 2019 Feb 14. PMID 30762420
- [Background] Drewniak D, Glassel A, Hodel M, Biller-Andorno N. Risks and Benefits of Web-Based Patient Narratives: Systematic Review. J Med Internet Res. 2020 Mar 26;22(3):e15772. doi: 10.2196/15772. PMID 32213468
- [Background] Inglis SC, Clark RA, McAlister FA, Stewart S, Cleland JG. Which components of heart failure programmes are effective? A systematic review and meta-analysis of the outcomes of structured telephone support or telemonitoring as the primary component of chronic heart failure management in 8323 patients: Abridged Cochrane Review. Eur J Heart Fail. 2011 Sep;13(9):1028-40. doi: 10.1093/eurjhf/hfr039. Epub 2011 Jul 6. PMID 21733889
- [Background] Clark RA, Inglis SC, McAlister FA, Cleland JG, Stewart S. Telemonitoring or structured telephone support programmes for patients with chronic heart failure: systematic review and meta-analysis. BMJ. 2007 May 5;334(7600):942. doi: 10.1136/bmj.39156.536968.55. Epub 2007 Apr 10. PMID 17426062
- [Background] Farahani MA, Mohammadi E, Ahmadi F, Mohammadi N. Factors influencing the patient education: A qualitative research. Iran J Nurs Midwifery Res. 2013 Mar;18(2):133-9. PMID 23983743
- [Background] Morton K, Beauchamp M, Prothero A, Joyce L, Saunders L, Spencer-Bowdage S, Dancy B, Pedlar C. The effectiveness of motivational interviewing for health behaviour change in primary care settings: a systematic review. Health Psychol Rev. 2015;9(2):205-23. doi: 10.1080/17437199.2014.882006. Epub 2014 Feb 12. PMID 26209209
- [Background] Anderson L, Brown JP, Clark AM, Dalal H, Rossau HK, Bridges C, Taylor RS. Patient education in the management of coronary heart disease. Cochrane Database Syst Rev. 2017 Jun 28;6(6):CD008895. doi: 10.1002/14651858.CD008895.pub3. PMID 28658719
- [Background] Ma C, Zhou W. Predictors of rehospitalization for community-dwelling older adults with chronic heart failure: A structural equation model. J Adv Nurs. 2020 Jun;76(6):1334-1344. doi: 10.1111/jan.14327. Epub 2020 Feb 26. PMID 32056280
- [Background] Ronksley PE, Sanmartin C, Campbell DJ, Weaver RG, Allan GM, McBrien KA, Tonelli M, Manns BJ, Hennessy D, Hemmelgarn BR. Perceived barriers to primary care among western Canadians with chronic conditions. Health Rep. 2014 Apr;25(4):3-10. PMID 24744042
- [Background] Jencks SF, Williams MV, Coleman EA. Rehospitalizations among patients in the Medicare fee-for-service program. N Engl J Med. 2009 Apr 2;360(14):1418-28. doi: 10.1056/NEJMsa0803563. PMID 19339721
- [Background] McCullough PA, Li S, Jurkovitz CT, Stevens LA, Wang C, Collins AJ, Chen SC, Norris KC, McFarlane SI, Johnson B, Shlipak MG, Obialo CI, Brown WW, Vassalotti JA, Whaley-Connell AT; Kidney Early Evaluation Program Investigators. CKD and cardiovascular disease in screened high-risk volunteer and general populations: the Kidney Early Evaluation Program (KEEP) and National Health and Nutrition Examination Survey (NHANES) 1999-2004. Am J Kidney Dis. 2008 Apr;51(4 Suppl 2):S38-45. doi: 10.1053/j.ajkd.2007.12.017. PMID 18359407
- [Background] Ndumele CE, Rangaswami J, Chow SL, Neeland IJ, Tuttle KR, Khan SS, Coresh J, Mathew RO, Baker-Smith CM, Carnethon MR, Despres JP, Ho JE, Joseph JJ, Kernan WN, Khera A, Kosiborod MN, Lekavich CL, Lewis EF, Lo KB, Ozkan B, Palaniappan LP, Patel SS, Pencina MJ, Powell-Wiley TM, Sperling LS, Virani SS, Wright JT, Rajgopal Singh R, Elkind MSV; American Heart Association. Cardiovascular-Kidney-Metabolic Health: A Presidential Advisory From the American Heart Association. Circulation. 2023 Nov 14;148(20):1606-1635. doi: 10.1161/CIR.0000000000001184. Epub 2023 Oct 9. Erratum In: Circulation. 2024 Mar 26;149(13):e1023. doi: 10.1161/CIR.0000000000001241. PMID 37807924